CLINICAL TRIAL: NCT04043624
Title: The Study of Perioperative Intravenous Infusion of Lidocaine on Postoperative Analgesia in Patients Undergoing Single-port Thoracoscopic
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-084
Record Dates: First submitted 2019-07-19; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Surgery
Keywords: single-port thoracoscopic surgery; lidocaine; postoperative pain; opioid
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): First group (lidocaine group) will include those who receive a intraoperative lidocaine infusion.Induction bolus dose of 1.5 mg/kg body weight ( 30 minutes before incision)followed by a continous lidocaine infusion of 2mg/kg/h，until 1 hours after skin closure.
  Interventions: Drug: Lidocaine
- Saline group (Placebo Comparator): The second group（saline group） will include those who receive a intraoperative placebo.The same dosage of saline was given according to the same method of administration in the lidocaine group.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Lidocaine — regimen of lidocaine administration of 1.5 mg/kg, IV bolus, followed by continuous infusion at 2 mg/kg/h
  Arms: Lidocaine group
Drug: Saline — IV bolus of saline, followed by continuous infusion of saline
  Arms: Saline group

SUMMARY:
The purpose of this study is to evaluate the effect of intravenous lidocaine infusion on pain and opioid dosage in patients undergoing single-port thoracoscopic surgery,and to evaluate the effects of perioperative catecholamine levels, extubation time, incidence of nausea and vomiting, patient satisfaction and hospital stay.

DETAILED DESCRIPTION:
The World Congress on Pain identified pain as the "fifth leading indicator of human life" after breathing, pulse, body temperature and blood pressure. Postoperative pain is an acute nociceptive pain caused by surgical trauma and is a complex stress response in the body, especially in 72 hours after surgery. Pain after thoracic surgery is a more severe type of surgery in various types of surgery.

Acute pain at the early stage of operation is not only an external signal of body injury, but also an independent factor inducing stress response and systemic inflammatory response syndrome (SIRS). Pain stimulus can also cause excessive release of catecholamine, damage of vascular endothelial cells and neutrophil aggregation, which can induce cytokine "waterfall" secretion. Stress, pain and inflammation induce and interact with each other, which seriously affects the early recovery of patients after operation. Timely and effective post-operative analgesia can not only alleviate patients'pain, but also avoid a series of stress reactions. It provides favorable conditions for the stability of patients' physiological function and recovery of their body after operation.

Although multimodal analgesia has largely replaced monotherapy with opioids, they are still the most commonly used drugs for postoperative pain. Lidocaine is an amide local anesthetic which when used intravenously demonstrates significant analgesic, anti-hyperalgesic and anti-inflammatory properties .

Intravenous infusion of lidocaine has a good effect on fibromyalgia, chronic neuropathic pain, opioid tolerance and other chronic pain, and can reduce postoperative acute pain. In the 1960s, Barlett et al. first published a study on the use of lidocaine intravenous infusion for postoperative analgesia.Since then, more and more researchers have begun to explore the use of lidocaine in the treatment of postoperative acute pain.In 2007, Kaba et al. selected patients who underwent colectomy as an experimental subject, and intravenously injected lidocaine during the perioperative period. The results showed that the pain of the experimental group was effectively relieved and the use of opioids was reduced. In 2008, Lauwick et al. used laparoscopic cholecystectomy as the experimental subject. The results showed that the dose of opioid analgesia in the lidocaine group was significantly lower than that in the control group, and the postoperative pain was effectively improved. In 2009, Yardeni et al. selected patients undergoing total hysterectomy as experimental subjects and intravenously injected lidocaine during the perioperative period. The results confirmed that the hemodynamics of the experimental group was more stable, the average dosage of anesthetics was reduced, and the pain was significantly improved.However, to date, there is no strong evidence for the effect of perioperative intravenous infusion of lidocaine in single-port thoracoscopic surgery, so we designed this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing single-port thoracoscopic with a left double lumen bronchial catheter
* Age ≧ 18 years old, ≦70 years old
* Temperature, white blood cells, and hemoglobin were normal before surgery
* Patient informed consent

Exclusion Criteria:

* Patients with a history of surgery within six months
* Patients with dysfunction of heart, liver, kidney, lung, pancreas or other important organs
* American Society of Anesthesiologists (ASA) physical Status classes ≧ Ⅲ
* Allergic to lidocaine
* Bradycardia (heart rate < 60 beats/min) or atrioventricular block
* Mental disorder
* Patients requiring a right double lumen bronchial catheter

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score | Immediately postoperation
  Using Visual Analogue Scales
Postoperative pain score | 1 hour postoperation
  Using Visual Analogue Scales
Postoperative pain score | 4 hours postoperation
  Using Visual Analogue Scales
Postoperative pain score | 8 hours postoperation
  Using Visual Analogue Scales
Postoperative pain score | 24 hours postoperation
  Using Visual Analogue Scales
Postoperative pain score | 48 hours postoperation
  Using Visual Analogue Scales

SECONDARY OUTCOMES:
Opioid requirement | Immediately postoperation
  The dosage of opioids was recorded
Opioid requirement | 1 hour postoperation
  The dosage of opioids was recorded
Opioid requirement | 4 hours postoperation
  The dosage of opioids was recorded
Opioid requirement | 8 hours postoperation
  The dosage of opioids was recorded
Opioid requirement | 24 hours postoperation
  The dosage of opioids was recorded
Opioid requirement | 48 hours postoperation
  The dosage of opioids was recorded
Pressing times of PCIA postoperation | 48 hours postoperation
  The pressing times of PCIA within 48 hours postoperation was recorded
Occurrence of nausea and/or vomiting | 48 hours postoperation
  The occurrence of nausea and vomiting within 48 hours postoperation was recorded
Blood level of adrenaline | before induction
  Perioperative blood level of adrenaline was recorded
Blood level of adrenaline | after incision
  Perioperative blood level of adrenaline was recorded
Blood level of adrenaline | immediately after extubation
  Perioperative blood level of adrenaline was recorded
Blood level of norepinephrine | before induction
  Perioperative blood level of norepinephrine was recorded
Blood level of norepinephrine | after incision
  Perioperative blood level of norepinephrine was recorded
Blood level of norepinephrine | immediately after extubation
  Perioperative blood level of norepinephrine was recorded
Blood level of adrenocortical | before induction
  Perioperative blood level of adrenocortical was recorded
Blood level of adrenocortical | after incision
  Perioperative blood level of adrenocortical was recorded
Blood level of adrenocortical | immediately after extubation
  Perioperative blood level of adrenocortical was recorded
Blood level of TNF-alpha | before induction
  Perioperative blood level of TNF-alpha was recorded
Blood level of TNF-alpha | after incision
  Perioperative blood level of TNF-alpha was recorded
Blood level of TNF-alpha | immediately after extubation
  Perioperative blood level of TNF-alpha was recorded
Blood level of IL-6 | before induction
  Perioperative blood level of IL-6 was recorded
Blood level of IL-6 | after incision
  Perioperative blood level of IL-6 was recorded
Blood level of IL-6 | immediately after extubation
  Perioperative blood level of IL-6 was recorded
Blood level of IL-10 | before induction
  Perioperative blood level of IL-10 was recorded
Blood level of IL-10 | after incision
  Perioperative blood level of IL-10 was recorded
Blood level of IL-10 | immediately after extubation
  Perioperative blood level of IL-10 was recorded
Duration of hospital stay | from day of surgery until day of discharge from hospital
  length of hospital stay (in days)

CONTACTS AND LOCATIONS:
Overall Officials: Congcong Chen, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Koppert W, Weigand M, Neumann F, Sittl R, Schuettler J, Schmelz M, Hering W. Perioperative intravenous lidocaine has preventive effects on postoperative pain and morphine consumption after major abdominal surgery. Anesth Analg. 2004 Apr;98(4):1050-1055. doi: 10.1213/01.ANE.0000104582.71710.EE. PMID 15041597
- [Background] Schafranski MD, Malucelli T, Machado F, Takeshi H, Kaiber F, Schmidt C, Harth F. Intravenous lidocaine for fibromyalgia syndrome: an open trial. Clin Rheumatol. 2009 Jul;28(7):853-5. doi: 10.1007/s10067-009-1137-8. Epub 2009 Mar 5. PMID 19263182
- [Background] Challapalli V, Tremont-Lukats IW, McNicol ED, Lau J, Carr DB. Systemic administration of local anesthetic agents to relieve neuropathic pain. Cochrane Database Syst Rev. 2005 Oct 19;2005(4):CD003345. doi: 10.1002/14651858.CD003345.pub2. PMID 16235318
- [Background] Buchanan DD, J MacIvor F. A role for intravenous lidocaine in severe cancer-related neuropathic pain at the end-of-life. Support Care Cancer. 2010 Jul;18(7):899-901. doi: 10.1007/s00520-010-0864-3. Epub 2010 Apr 29. PMID 20429016
- [Background] Sharma S, Rajagopal MR, Palat G, Singh C, Haji AG, Jain D. A phase II pilot study to evaluate use of intravenous lidocaine for opioid-refractory pain in cancer patients. J Pain Symptom Manage. 2009 Jan;37(1):85-93. doi: 10.1016/j.jpainsymman.2007.12.023. Epub 2008 Jul 2. PMID 18599258
- [Background] Lauwick S, Kim DJ, Michelagnoli G, Mistraletti G, Feldman L, Fried G, Carli F. Intraoperative infusion of lidocaine reduces postoperative fentanyl requirements in patients undergoing laparoscopic cholecystectomy. Can J Anaesth. 2008 Nov;55(11):754-60. doi: 10.1007/BF03016348. PMID 19138915
- [Background] Kaba A, Laurent SR, Detroz BJ, Sessler DI, Durieux ME, Lamy ML, Joris JL. Intravenous lidocaine infusion facilitates acute rehabilitation after laparoscopic colectomy. Anesthesiology. 2007 Jan;106(1):11-8; discussion 5-6. doi: 10.1097/00000542-200701000-00007. PMID 17197840
- [Background] Yardeni IZ, Beilin B, Mayburd E, Levinson Y, Bessler H. The effect of perioperative intravenous lidocaine on postoperative pain and immune function. Anesth Analg. 2009 Nov;109(5):1464-9. doi: 10.1213/ANE.0b013e3181bab1bd. PMID 19843784
- [Background] Eriksson AS, Sinclair R, Cassuto J, Thomsen P. Influence of lidocaine on leukocyte function in the surgical wound. Anesthesiology. 1992 Jul;77(1):74-8. doi: 10.1097/00000542-199207000-00011. PMID 1610012
- [Background] Feng G, Liu S, Wang GL, Liu GJ. Lidocaine attenuates lipopolysaccharide-induced acute lung injury through inhibiting NF-kappaB activation. Pharmacology. 2008;81(1):32-40. doi: 10.1159/000107792. Epub 2007 Sep 4. PMID 17785997